CLINICAL TRIAL: NCT06807541
Title: The Effect of a Group Exercise Intervention on Balance in People With Knee Osteoarthritis: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Fraser Valley (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101716
Record Dates: First submitted 2025-01-20; First posted 2025-02-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; balance; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise program (Experimental): Twice weekly exercise classes, for 12 weeks
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — 45 minute exercise classes. Twice per week for 12 weeks.

SUMMARY:
In this study, the investigators want to find out if a 12-week exercise program improves balance in people with knee osteoarthritis.

This study will involve two visits to the School of Kinesiology at the University of the Fraser Valley (Chilliwack campus). Each visit will last approximately one hour. Participants will be asked to fill out questionnaires and complete a balance test. In between visits, participants will complete 12 weeks of an exercise program specifically designed for adults with osteoarthritis. Participants will do the exercise classes twice per week. Classes can be done in person or at home

Each exercise class is 45-minutes long and consists of flexibility, strength, and coordination exercises. In each class there are options to either increase or decrease the intensity of each exercise to cater to varying fitness levels and fluctuating symptoms. Each exercise has an assisted (using a chair for balance), body weight, and resisted (weight or exercise tubing) option. Participants will fill out an exercise diary each week to let the investigators know what days they did the exercise classes, and whether they experienced any changes in their knee osteoarthritis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Medial compartment knee osteoarthritis, diagnosed from a physician or meeting the American College of Rheumatology Clinical Classification Criteria for Osteoarthritis of the knee
* Pass the Get Active Questionnaire to ensure that they are safe to begin an exercise program

Exclusion Criteria:

i) severe knee trauma, knee surgery, or intraarticular knee joint injections in the previous six months ii) active synovitis iii) concurrent neurological (i.e. Parkinson's disease, Alzheimer's dementia, or polyneuropathy), endocrine (i.e., diabetes mellitus) and/or vestibular disorders which may affect balance iv) chronic disease that may put them at risk during the exercise classes (i.e., history of heart failure, stroke, chronic obstructive lung disease) v) uncorrected visual impairment which may affect balance vi) an inflammatory rheumatic disease (i.e., rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, and chronic reactive arthritis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-06-19 (Estimated)

PRIMARY OUTCOMES:
Balance- Community Balance and Mobility Scale | From enrolment until the end of the treatment at 12 weeks.
  Community Balance and Mobility Scale- scaled from 0 to 96, where higher scores indicate higher balance (better outcome).

SECONDARY OUTCOMES:
Symptoms- Western Ontario and McMaster University Osteoarthritis Index | From enrolment until the end of the treatment at 12 weeks.
  Western Ontario and McMaster University (WOMAC) Osteoarthritis Index- Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status.
Symptoms- Oxford Knee Score | From enrolment until the end of the treatment at 12 weeks.
  The Oxford Knee Score is scored from 0-48, where higher scores are a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Hatfield, PhD, Principal Investigator — University of the Fraser Valley
Locations (1):
- University of the Fraser Valley, Chilliwack, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified pre and post intervention data (age, sex, height, mass, WOMAC and Oxford Knee Score scores, and Community Balance and Mobility Scores) will be shared on reasonable request.
Supporting Information: Study Protocol
Time Frame: Available from August 2025 until August 2034
Access Criteria: Data will be shared with other researchers at academic institutions. A proposal that describes planned analyses must be submitted and a data sharing agreement must be signed. Proposals may be submitted to the primary investigator for review.